CLINICAL TRIAL: NCT02479451
Title: Helping Olfaction and Nutrition On Renal Replacement
Acronym: HONORR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sagar U. Nigwekar, MD, MMSc, Assistant in Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P001231
Record Dates: First submitted 2015-06-18; First posted 2015-06-24 (Estimated); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-11

CONDITIONS: End Stage Renal Disease; Olfactory Disorders
Keywords: End stage renal disease; Olfaction; Dialysis; Hemodialysis; Malnutrition
MeSH Terms: conditions — Kidney Failure, Chronic; Anosmia; Malnutrition | interventions — Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nasal theophylline (Experimental): 20 μg intranasal theophylline (theophylline methylpropyl paraben in a 0.4-mL saline solution) once daily (in the morning) into each naris for a total of 6 weeks
  Interventions: Drug: Theophylline

INTERVENTIONS:
Drug: Theophylline — The study medication will be provided by Foundation Care.

SUMMARY:
This clinical trial examines whether nasal theophylline administration can improve olfaction and nutrition in hemodialysis patients.

DETAILED DESCRIPTION:
Malnutrition and cachexia are prevalent in end stage renal disease (ESRD) patients and are associated with increased morbidity and mortality. Food aversion is a major contributor to anorexia and malnutrition in ESRD and it also impacts the quality of life. Olfactory dysfunction has been shown to contribute to food aversion in ESRD patients. Since up to 80% of a meal's flavor is attributed to olfactory input, loss or alteration of smell leads to loss or alteration of taste in ESRD patients and at present there are no effective therapies to treat smell and/or taste disorders in ESRD patients.

In patients with other causes of olfactory dysfunction such as congenital hyposmia and traumatic brain injury, intranasal theophylline has been shown to be effective in improving olfactory defects via increasing nasal mucus levels of cAMP and cGMP, second messengers critical for optimal smell sensation. However, the efficacy of nasal theophylline to improve olfaction in ESRD patients has not been investigated and the effects of nasal theophylline treatment on the nutritional parameters are unknown in ESRD patients.

Aim: To examine the efficacy and safety of nasal theophylline treatment to improve olfaction and nutrition in ESRD patients

Hypothesis: Nasal theophylline treatment improves olfaction and nutrition in ESRD patients with olfactory defects by via increasing intracellular cAMP and cGMP levels.

A previous pilot clinical trial demonstrated that intranasal theophylline is safe and effective in improving olfactory deficits in congenital hyposmia and traumatic brain injury, however, it has not been examined in ESRD patients. The investigators will conduct a pilot single arm open-label clinical trial (n=20) of 6 weeks duration to examine the efficacy and safety of nasal theophylline in hemodialysis-dependent ESRD patients with olfactory defects. The investigators will examine whether nasal theophylline improves olfaction and nutritional status in trial participants.

ELIGIBILITY:
Inclusion Criteria:

* ESRD requiring chronic outpatient hemodialysis
* Able to provide written consent
* Defects in smell identification and/or smell threshold detection as measured by "Scratch-and-sniff" University of Pennsylvania Smell Identification Test (UPSIT) and Smell Threshold Test

Exclusion Criteria:

* Prior allergic reaction to theophylline
* Patients currently treated with theophylline for clinical indication
* Pregnancy or lactation
* ESRD patients on peritoneal dialysis
* Patients hospitalized at the time of study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2022-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sagar U Nigwekar, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Henkin RI, Velicu I, Schmidt L. An open-label controlled trial of theophylline for treatment of patients with hyposmia. Am J Med Sci. 2009 Jun;337(6):396-406. doi: 10.1097/MAJ.0b013e3181914a97. PMID 19359985
- [Background] Henkin RI, Schultz M, Minnick-Poppe L. Intranasal theophylline treatment of hyposmia and hypogeusia: a pilot study. Arch Otolaryngol Head Neck Surg. 2012 Nov;138(11):1064-70. doi: 10.1001/2013.jamaoto.342. PMID 23165381

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Theophylline
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All adult patients with ESRD treated with HD
Arm/Group | Nasal Theophylline
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 55 [45 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
ESRD [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Smell Identification Test Score at 6 Weeks
Description: Smell identification test is a validated 40-item scratch and sniff smell identification test that was administered by study investigators. Scores on this test scale range between 0 (minimum) to 40 (maximum). Higher score indicates better ability for smell identification. Total scores are reported on this scale (no sub-scales). The unit is score on this scale.
Time Frame: Baseline and every 2 weeks for 6 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Nasal Theophylline
Number analyzed (Participants) | 7
units on a scale | 4 (2)

2. Primary Outcome: Change From Baseline in Smell Threshold Test Score at 6 Weeks
Description: This test determined the lowest concentration of an odor compound that is perceivable by study participants. Scores on this test scale range between -2 and -10.
  Higher score indicates higher smell detection threshold (i.e. worse ability to smell). Total scores are reported on this scale (no sub-scales). The unit is score on this scale.
Time Frame: Baseline and every 2 weeks for 6 weeks
Measure: Mean (Standard Error); unit: change in score on the scale
Arm/Group | Nasal Theophylline
Number analyzed (Participants) | 7
change in score on the scale | -1 (2)

3. Secondary Outcome: Change From Baseline in Plasma Theophylline Level at 6 Weeks
Description: Plasma levels of theophylline were measured using fluorescence polarization technique. Minimum level will be 0 microgram/mL and maximum assay limit is 40 microgram/mL. Higher levels indicate increased systemic exposure to theophylline. Units on scale are microgram/mL.
Time Frame: Baseline and every 2 weeks for 6 weeks
Population: Serum theophylline levels assessed at every follow-up were undetectable throughout the study period in all participants.
Measure: Mean (Standard Deviation); unit: microgram/mL
Arm/Group | Nasal Theophylline
Number analyzed (Participants) | 7
microgram/mL | 0 (0)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Nasal Theophylline
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT02479451/Prot_000.pdf